CLINICAL TRIAL: NCT02171533
Title: Relative Bioavailability of Single Oral Doses of 150 mg Dabigatran Etexilate With or Without Oral Administration of Verapamil in Two Different Dosages (240 mg and 480 mg Daily) (Open-label, Fixed-sequence Design), and Relative Bioavailability of Single Oral Doses of 150 mg Dabigatran Etexilate Given With or Without Single Oral Doses of 120 mg (IR) or 240 mg (ER) of Verapamil Administered at Different Time Points Relative to Dabigatran Etexilate Dosing in Healthy Male and Female Volunteers (Open-label, Randomised, Five-way Crossover Design, Phase I Study)
Brief Title: Relative Bioavailability of Single Oral Doses of Dabigatran Etexilate With or Without Oral Administration of Verapamil in Two Different Dosages in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.74
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Verapamil

ARMS (2):
- Fixed sequence (Experimental): Treatments will be given in a fixed sequence
  Interventions: Drug: dabigatran; Drug: Verapamil
- Crossover (Experimental): Treatments will be given in randomized sequences
  Interventions: Drug: dabigatran; Drug: Verapamil; Drug: Verapamil ER

INTERVENTIONS:
Drug: dabigatran
Drug: Verapamil
Drug: Verapamil ER
  Arms: Crossover

SUMMARY:
To investigate whether and to what extent the P-glycoprotein inhibitor (P-gp) verapamil affects the pharmacokinetic parameters of dabigatran with verapamil given at different dosages, in different formulations (immediate release (IR) and extended release (ER)), and in different intervals in relation to the dabigatran dose.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age ≥18 and ≤55 years
3. Body mass index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Pulse rate below 50 bpm and or systolic blood pressure <90 mm Hg at screening. ECG: PR >170 ms (Part 1), AV block ≥1st degree (Part 2) at screening
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within four weeks prior to administration or during the trial, especially intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, cumarin etc.
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (more than 15 cigarettes or 3 cigars or 3 pipes per day)
12. Alcohol abuse (more than 60 g/day for men and more than 40 g/day for women)
13. Drug abuse
14. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
15. Excessive physical activities (within one week prior to administration or during the trial)
16. Any laboratory value outside the reference range that is of clinical relevance
17. Planned surgeries within four weeks following the end-of study examination
18. The subject is not able to understand and comply with protocol requirements, instructions, protocol-stated restrictions and dietary regimen of study centre

    For male subjects:
19. Male subjects who do not agree to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post study medical. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)

    For female subjects:
20. Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
21. No adequate contraception during the study and until 1 month of study completion, i.e. implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females, who have not a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
22. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of total dabigatran over the time interval from 0 extrapolated to infinity) | up to 107 hours
Cmax (maximum measured concentration of total dabigatran) | up to 107 hours

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of free dabigatran over the time interval from 0 extrapolated to infinity) | up to 107 hours
Cmax (maximum measured concentration of free dabigatran) | up to 107 hours
AUC0-infinity (area under the concentration-time curve of verapamil over the time interval from 0 extrapolated to infinity) | up to 107 hours
Cmax (maximum measured concentration of verapamil) | up to 107 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 107 hours
AUC0-24 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h after the administration) | up to 107 hours
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 107 hours
λz (terminal rate constant in plasma) | up to 107 hours
t1/2 (terminal half-life of the analyte in plasma) | up to 107 hours
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 107 hours
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 107 hours
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 107 hours
AUCτ,ss (area under the concentration-time curve of verapamil within the uniform dosing interval τ) | up to 107 hours
AUC0-tz,ss (area under the concentration-time curve of verapamil from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ) | up to 107 hours
Cmax,ss (maximum concentration of verapamil at steady state) | up to 107 hours
tz,ss (time of last measureable concentration of verapamil within the dosing interval τ at steady state) | up to 107 hours
tmax,ss (time from last dosing to the maximum concentration of verapamil at steady state on day 4) | up to 107 hours
CL/F,ss (apparent clearance of verapamil at steady state after extravascular multiple dose administration) | up to 107 hours
Cmin,ss (minimum measured concentration of verapamil at steady state over a uniform dosing interval τ) | up to 107 hours
tmin,ss (time from last dosing to the minimum concentration of verapamil at steady state over a uniform dosing interval τ) | up to 107 hours
Cpre,ss (predose concentration of verapamil at steady state immediately before administration of the next dose) | up to 107 hours
Cavg (Average concentration of verapamil at steady state) | up to 107 hours
MRTpo,ss (mean residence time of verapamil in the body at steady state after oral administration) | up to 107 hours
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration) | up to 107 hours
Ae0-24 (amount of dabigatran that is eliminated in urine from the time interval 0-24h) | up to 107 hours
fe0-24 (fraction of administered drug excreted unchanged in urine from time point 0- 24h) | up to 107 hours
CLR0-24 (renal clearance of dabigatran from the time point 0 until the time point 24h ) | up to 107 hours
AUEC0-24 (area under the effect curve) | up to 107 hours
  for ecarin clotting time and thrombin time
ERmax (maximum effect ratio) | up to 107 hours
  for ecarin clotting time and thrombin time
Occurence of Adverse Events | within 5 days after last drug administration
Assessment of Tolerability by investigator | within 5 days after last drug administration